CLINICAL TRIAL: NCT00147043
Title: Adult Stem Therapy for Patients With Liver Insufficiency
Brief Title: Adult Stem Cell Therapy in Liver Insufficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004/6746
Record Dates: First submitted 2005-09-05; First posted 2005-09-07 (Estimated); Results first posted 2019-10-03 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Liver Cirrhosis
Keywords: Adult stem cells; Liver disease; CD34 positive cells
MeSH Terms: conditions — Liver Cirrhosis; Liver Diseases | interventions — Leukapheresis

STUDY DESIGN:
Intervention Model Description: Autologous stem cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous Stem Cells (Experimental)
  Interventions: Procedure: Leukapheresis; Procedure: Infusion of stem cells via image guided scan

INTERVENTIONS:
Procedure: Leukapheresis
Procedure: Infusion of stem cells via image guided scan

SUMMARY:
In order to determine the clinical application potential of adult stem cells we propose to investigate the safety and toxicity of infusing adult stem cells in the hepatic artery or portal vein of five patients with chronic liver insufficiency and to identify any clinical benefit if such occurs.

Objectives:

1. To assess safety and treatment related toxicities
2. To determine clinical benefit or deterioration by monitoring changes in liver function

DETAILED DESCRIPTION:
The liver in an adult healthy body maintains a balance between cell gain and cell loss. Though normally proliferatively quiescent, hepatocyte loss such as that caused by partial hepatectomy, uncomplicated by virus infection or inflammation, invokes a rapid regenerative response to restore liver mass. This restoration of moderate cell loss and 'wear and tear' renewal is largely achieved by hepatocyte self-replication. More severe liver injury can activate a potential stem cell compartment located within the intrahepatic biliary tree, giving rise to cords of bipotential, so-called, oval cells within the lobules that can differentiate into hepatocytes and biliary epithelial cells. A third population of stem cells with hepatic potential reside in the bone marrow; these haematopoietic stem cells can contribute to the albeit low renewal rate of hepatocytes, make a more significant contribution to regeneration and even completely restore normal function in a murine model of hereditary tyrosinaemia.

A recent abstract has suggested that an astonishingly high number of bone marrow cells (~25% of liver parenchyma occupied by bone marrow-derived cells) will engraft and differentiate into hepatocytes in a model of cirrhosis in the mouse when injected intravenously. More importantly, this bone marrow infusion resulted in significant improvements in liver function (serum albumin) within the cirrhotic animals.

This is a safety and toxicity study in five patients with chronic liver disease. Each will receive autologous stem cells 10 to the sixth cells via the hepatic artery or portal vein under image guided scanning. Patients will be followed for a total of 60 days.

ELIGIBILITY:
Inclusion Criteria:

- Male or female aged from 20 years to 65 years Evidence of chronic liver failure Abnormal serum albumin and/or bilirubin and/or prothrombin time Unsuitable for liver transplantation WHO performance status <2 Women of childbearing potential may be included but must use a reliable and appropriate contraceptive method Life expectancy of at least three months Ability to give informed consent

Exclusion Criteria:

- Patients aged below 20 years or above 65 years Pregnant or lactating women Patients with recent recurrent gastrointestinal bleeding Spontaneous bacterial peritonitis Evidence of active infection HIV infection Patients unable to give informed consent

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nagy Habib, ChM FRCS, Principal Investigator — Imperial College London
Locations (1):
- Hammersmith Hospitals NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gordon MY, Levicar N, Pai M, Bachellier P, Dimarakis I, Al-Allaf F, M'Hamdi H, Thalji T, Welsh JP, Marley SB, Davies J, Dazzi F, Marelli-Berg F, Tait P, Playford R, Jiao L, Jensen S, Nicholls JP, Ayav A, Nohandani M, Farzaneh F, Gaken J, Dodge R, Alison M, Apperley JF, Lechler R, Habib NA. Characterization and clinical application of human CD34+ stem/progenitor cell populations mobilized into the blood by granulocyte colony-stimulating factor. Stem Cells. 2006 Jul;24(7):1822-30. doi: 10.1634/stemcells.2005-0629. Epub 2006 Mar 23. PMID 16556705

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were sequentially recruited to the study from January 2005 to June 2005
Groups:
- Autologous Stem Cells: Pre-treatment with Granulocyte-Colony Stimulating Factor (G-CSF) to mobilise CD34+ cells Leukapheresis procedure to extract mobilised CD34+ cells Cultured CD34+ cells administered via hepatic artery of portal vein
Period: Overall Study
Arm/Group | Autologous Stem Cells
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Autologous Stem Cells: Male or female aged from 20 years to 65 years with evidence of chronic liver failure, abnormal serum albumin and/or bilirubin and/or prothrombin time
Arm/Group | Autologous Stem Cells
Number analyzed (Participants) | 5
Age, Continuous [Mean (Full Range); unit: years] — Mean Age
  years | 49 [41 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Gender: Female | 1
  Gender: Male | 4
Region of Enrollment [Number; unit: participants]
  United Kingdom | 5
Count of Participants [Count of Participants; unit: Participants] | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events Related to Injection
Description: Incidence of serious adverse event related to injection with the study participants
Time Frame: Day 1 to Day 60
Measure: Count of Participants; unit: Participants
Groups:
- Autologous Stem Cells: Male of Female participants aged from 20-65 years old with chronic liver failure Abnormal liver function Abnormal serum albumin and/or bilirubin and/or prothrombin time Unsuitable for liver transplantation WHO Performance status <2 Women of childbearing potential may be included but must use a reliable and appropriate contraceptive method Life expectancy of at least 3 monthsAbility to give informed consent
Arm/Group | Autologous Stem Cells
Number analyzed (Participants) | 5
Participants | 0

2. Secondary Outcome: Improvement in Liver Function
Description: Number of participant that have liver function improvement in liver function
Time Frame: Day 1 to Day 60
Measure: Count of Participants; unit: Participants
Groups:
- Autologous Stem Cells: Leukapheresis
  Infusion of stem cells via image guided scan
Arm/Group | Autologous Stem Cells
Number analyzed (Participants) | 5
Participants | 5

ADVERSE EVENTS:
Time Frame: 60 days
Groups:
- Autologous Stem Cells: Male of Female participants aged from 20-65 years old with chronic liver failure, abnormal liver function, abnormal serum albumin and/or bilirubin and/or prothrombin time
Arm/Group | Autologous Stem Cells
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
The study was limited to 5 participants, which is an insufficient number to determine true benefit. A larger Phase I/II should be undertaken to determine benefit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes